CLINICAL TRIAL: NCT01903161
Title: Effect of Delayed Remote Ischemic Preconditioning on Myocardial Injury in Patients Undergoing Cardiac Valve Replacement Surgery
Brief Title: Effect of Delayed Remote Ischemic Preconditioning on Myocardial Injury
Acronym: RIPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: delayed RIPC
Record Dates: First submitted 2013-07-01; First posted 2013-07-19 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Myocardial Injury
Keywords: delayed remote ischemic preconditioning; troponin; valve replacement surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- delayed remote ischemic preconditioning (Experimental): applying pneumatic cuff on upper extremity (5 minutes cycles of limb ischemia and reperfusion with pneumatic cuff up to 200 mmHg repeated by four times)
  Interventions: Procedure: delayed remote ischemic preconditioning
- control (Placebo Comparator): All the procedures were the same in the control group, except for the fact that the three-way stopcock between the pneumatic cuff and the cuff inflator was opened and therefore the cuff pressure did not increase.
  Interventions: Procedure: control

INTERVENTIONS:
Procedure: delayed remote ischemic preconditioning — In the delayed RIPC group, RIPC is performed 24-48 hr before surgery by 5 minutes limb ischemia and reperfusion with pneumatic cuff up to 200 mmHg repeated by four times.
  Arms: delayed remote ischemic preconditioning
Procedure: control — In the control group, all the procedures were the same with delayed RIPC group, except for the fact that the three-way stopcock between the pneumatic cuff and the cuff inflator was opened and therefore the cuff pressure did not increase.
  Arms: control

SUMMARY:
The purpose of this study is to evaluate delayed myocardial protective effect of RIPC in patients undergoing cardiac valve replacement surgery.

DETAILED DESCRIPTION:
Ischemic preconditioning is one of the strategies that can reduce perioperative myocardial injury. It is a concept that briefly induced ischemia and reperfusion before the myocardial injury can reduce the myocardial injury. But it is difficult to apply ischemic preconditioning in operative field, because cross-clamping of aorta or coronary artery is difficult and invasive. Afterward concept of remote ischemic preconditioning(RIPC) has introduced that ischemia of remote organs like kidneys, skeletal muscles can reduce distant myocardial injury.

It is known that myocardial protective effect of ischemic preconditioning have biphasic pattern. Early protective effect wanes after a few hours, then recurs after 24-48 hours, and can persist for up to 3-4 days. It is called second window of preconditioning or delayed ischemic preconditioning. Delayed ischemic preconditioning is similar to early ischemic preconditioning in mechanism but it is different that it produces protein that can mediate myocardial protection effect.

Unlike ischemic preconditioning, it is little known about delayed effect of RIPC. RIPC can be done by applying compression cuff on upper or lower extremities and it is noninvasive and easy to deliver compared to ischemic preconditioning that is done by aorta or coronary artery clamping.

Delayed ischemic preconditioning is performed one day before the surgery, and it is safe and easy to apply RIPC in a clinical setting. And in this study investigators are going to evaluate cardioprotective effect of delayed RIPC. Myocardial injury can be predicted by elevation of cardiac enzyme. Investigators are going to perform RIPC one day before the valve replacement surgery and compare troponin I with control group to assess cardioprotective effect of delayed RIPC.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 80 years of adult patient undergoing cardiac valve surgery

Exclusion Criteria:

* Patient who did not agree to the study
* Emergency operation
* Using inotropics, mechanical assisting device
* Severe liver disease (>Child class II )
* Severe renal disease (Renal replacement therapy)
* left ventricular ejection fraction < 30%
* Co-operation of major surgery (Carotid endarterectomy )
* Oral hypoglycemic agent (Sulfonylurea, Glibenclamide)
* peripheral vascular disease affecting upper extremity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Troponin I change | before induction of anesthesia, postoperative 1, 6, 12, 24, 48, 72 hours

SECONDARY OUTCOMES:
serum creatinine changes | before induction of anesthesia, postoperative 1, 3, 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Deok Man Hong, M.D., Ph. D., Study Director — Seoul National University Hospital; Tae Kyong Kim, M.D., Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea